CLINICAL TRIAL: NCT02091076
Title: Efficacy and Safety of Wound Dressing Containing Silk Fibroin With Bioactive Coating Layer Versus Medicated Paraffin Gauze Dressing in the Treatment of Split-thickness Skin Graft Donor Sites
Brief Title: Efficacy and Safety of Silk Fibroin With Bioactive Coating Layer Dressing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Chula-53-1
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Late Complication From Skin Graft; Infection of Skin Donor Site; Impaired Wound Healing; Pain, Intractable
Keywords: Silk fibroin with bioactive coating layer dressing; Wound healing; Skin graft donor
MeSH Terms: conditions — Pain, Intractable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silk with bioactive coated dressing (Experimental): Silk fibroin coated with bioactive layer, apply once only
  Interventions: Device: Silk fibroin with bioactive coating layer dressing
- Control (Active Comparator): Bactigras wound dressing, apply once only
  Interventions: Device: Bactigras wound dressing

INTERVENTIONS:
Device: Silk fibroin with bioactive coating layer dressing
  Arms: Silk with bioactive coated dressing
Device: Bactigras wound dressing
  Arms: Control

SUMMARY:
A split-thickness skin graft (STSG) is used for a large wounds or wounds that cannot be closed by primary and secondary wound closure. Accelerated re-epithelialization rate and minimizing pain and infection are main goals of donor care. Traditionally dressings are inexpensive but adhere to the wound surface and cannot absorb exudates. Thus, we have developed a new biomaterial based on Thai silk for wound dressing application. Silk fibroin and silk sericin were selected to produce wound dressing in this study. The objective of this study is to compare wound dressing containing silk fibroin with bioactive coating layer with standard dressing (medicated paraffin gauze dressing; Bactigras®), with regard to healing time, patients' pain intensity, skin's transepidermal water loss after healing and evidence of infection in the treatment of split-thickness skin graft donor sites. The study design is a randomized, controlled, self paired clinical trial. Patients age 18 to 60 years and undergo STSG at thigh in Department of Surgery, King Chulalongkorn Memorial Hospital will be recruited in the study. The exclusion criteria are donor sites other than thigh area or located at high risk of infection. Patients who are immunocompromised or diabetes mellitus or psychiatric disorders or low serum albumin level (less than 3.0 g/dL) or known allergic to SS or SF or paraffin or chlorhexidine acetate are also excluded. All subjects sign the informed consents after discussion the protocol, benefits and risks. The donor site will be divided into two equal halves, each site will be randomized to receive the tested material or the medicated paraffin gauze dressing. The donor site wounds will be observed daily. The dressings will not be changed, except when they are fully soaked with exudates and easily fell off or any sign of infection. Healing time will be recorded when the dressing separate completely from the donor site, no exudates and no pain when the donor site is exposed to air. The patient's pain level will be evaluated with the visual analogue scale and the donor site wounds will be observed daily for signs of infection. On the day of the wound is recorded for healing time and 1 weeks, 1, 2, 3, 4 and 5 months after that, the skin barrier function (TEWL) of each site will be measured using a Tewameter. Blood sample will be collected from patients pre- and postoperatively (within day 3) for hepatic and renal function analysis.

DETAILED DESCRIPTION:
1. To compare the healing times of the split-thickness skin graft donor site under wound dressing containing silk fibroin woven fabric with bioactive coating layer and medicated paraffin gauze dressing.
2. To compare the patients' pain levels of the split-thickness skin graft donor site under wound dressing containing silk fibroin woven fabric with bioactive coating layer and medicated paraffin gauze dressing.
3. To compare the chance of infections of the split-thickness skin graft donor site under wound dressing containing silk fibroin woven fabric with bioactive coating layer and medicated paraffin gauze dressing.
4. To determine the complications with the use of wound dressing containing silk fibroin woven fabric with bioactive coating layer.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 to 60 years.
* Patients have to undergo a split thickness skin graft.
* The donor sites of split-thickness skin graft locate on the thigh.
* Patients consent to participate in this study.

Exclusion Criteria:

* Donor sites are anywhere else than the thigh area.
* Patients are allergic to silk sericin or silk fibroin or paraffin or chlorhexidine acetate.
* There is a risk of transferring an infection from a nearby infected area to donor site such as acute burn patients.
* Immunocompromised patients such as with acquired immunodeficiency syndrome (AIDS) and renal failure.
* Patients with diabetes mellitus.
* Patients with low serum albumin level (less than 3.0 g/dL)
* Patients have psychiatric disorders or patients with physical disabilities that hinders collaboration.
* Patients who do not comply with the study protocol.
* Pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of of wound dressing containing silk fibroin with bioactive coating layer dressing in the treatment of split-thickness skin graft donor sites | Within 14 days after operation
  Time for complete epithalization is duration between finishing surgical procedure and the dressing spontaneously peeling off from donor sites without causing pain. The wounds completely close and without fluid leakage and are able to exposed to the environment without pain. This duration should not exceed than 14 days.

SECONDARY OUTCOMES:
Clinical safety of wound dressing containing silk fibroin with bioactive coating layer dressing in the treatment of split-thickness skin graft donor sites | Within 14 days after operation
  Percentage of wound infection

OTHER OUTCOMES:
Clinical safety of wound dressing containing silk fibroin with bioactive coating layer dressing in the treatment of split-thickness skin graft donor sites | Within 14 days after operation
  Pain assessment is evaluated by patients themselves
Clinical safety of wound dressing containing silk fibroin with bioactive coating layer dressing in the treatment of split-thickness skin graft donor sites | Within 14 days after operation
  Laboratory measurement such as CBC, blood glucose, electrolyte, hepatic and renal function will be analyzed to find any changes or any systemic effect after treatment
Clinical safety of wound dressing containing silk fibroin with bioactive coating layer dressing in the treatment of split-thickness skin graft donor sites | Within 14 days after operation
  Transepidermal water loss (TEWL) measurement will be analyzed to find improvement in the rate of reestablishment of skin barrier function

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn Hospital, Bangkok, Bangkok, Thailand